CLINICAL TRIAL: NCT02172911
Title: Phase I/IIA, Open-Label, Safety, Tolerability, and Immunogenicity Study of INO-3112 Delivered by Electroporation (EP) in Women With Cervical Cancer After Chemoradiation for Newly Diagnosed Disease or Therapy for Recurrent and/or Persistent Disease
Brief Title: A Study of INO-3112 DNA Vaccine With Electroporation in Participants With Cervical Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Inovio Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HPV-004
Record Dates: First submitted 2014-05-18; First posted 2014-06-24 (Estimated); Results first posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Cervical Cancer
Keywords: Cervical cancer; Papillomavirus; Chemoradiation; Recurrent cervical cancer; Persistent cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — MEDI0457; VGX-3100; rocakinogene sifuplasmid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Cohort I: INO-3112: Curative Intent (Experimental): Cohort I included participants with biopsy-proven, stage IB-IVB inoperable, newly diagnosed invasive cervical carcinoma associated with HPV-16 and/or HPV-18 treated with standard chemoradiation therapy with curative intent. Participants received a 4-dose series of 1.1 mL IM injection of INO-3112 followed immediately by EP with CELLECTRA™-5P.
  Interventions: Biological: INO-3112; Device: CELLECTRA™-5P
- Cohort II: INO-3112: Salvage Therapy (Experimental): Cohort II included participants with persistent and/or recurrent cervical carcinoma associated with HPV-16 and/or HPV-18 who had been treated with salvage therapy (chemotherapy and/or radiation therapy). Participants received a 4-dose series of 1.1 mL IM injection of INO-3112 followed immediately by EP with CELLECTRA™-5P.
  Interventions: Biological: INO-3112; Device: CELLECTRA™-5P

INTERVENTIONS:
Biological: INO-3112 — 1.1 mL intramuscular (IM) injection of INO-3112 (VGX-3100 + INO-9012) was administered followed immediately by electroporation (EP) with CELLECTRA™-5P on Day 0, Week 4, Week 8, and Week 12.
  Other Names: VGX-3100; INO-9012
Device: CELLECTRA™-5P — CELLECTRA™-5P was used for EP following IM delivery of INO-3112 on Day 0, Week 4, Week 8, and Week 12.

SUMMARY:
This is an open-label study to evaluate the safety, tolerability, and immunogenicity of INO-3112 DNA vaccines delivered by electroporation (EP) to female participants with HPV-16 and/or 18-positive cervical carcinoma.

DETAILED DESCRIPTION:
This is a Phase I/IIa, open-label study to evaluate the safety, tolerability, and immunogenicity of INO-3112 [VGX-3100 and INO-9012] delivered intramuscularly by electroporation in approximately 30 female participants with biopsy-proven, Stage IB-IVB inoperable invasive cervical carcinoma associated with HPV 16 and/or 18 who have completed treatment with standard chemoradiation therapy with curative intent (Cohort I) or in participants with persistent and/or recurrent cervical cancer associated with HPV 16 and/or 18 following salvage therapy (Cohort II).

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Histological diagnosis of squamous cell carcinoma, adenocarcinoma or adenosquamous cell carcinoma of the cervix. Not accepted are small cell, clear cell and other rare variants of the classical adenocarcinoma.
3. Histologically confirmed, Stage IB-IVB, invasive cervical carcinoma associated with HPV 16 and/or 18 and meet the following eligibility criteria for either Cohort 1 or Cohort 2.

   1. Cohort 1

      * Newly diagnosed inoperable cervical cancer treated with chemoradiation therapy with curative intent and life expectancy of at least 12 months as assessed by the investigator
      * No CNS/spinal metastases
      * Able to initiate study treatment within 2 weeks of completion of last chemoradiation treatment
   2. Cohort 2

      * Persistent and/or recurrent cervical cancer
      * No CNS/spinal metastases
      * Able to initiate study treatment at least 2 weeks but no more than 4 weeks after completion of salvage therapy
      * Life expectancy of at least 12 months as assessed by the investigator
4. Electrocardiogram (ECG) with no clinically significant findings.
5. Chemistry, liver function tests, renal function, total CPK and hematology lab results must be ≤ Grade 1 at the time of screening.
6. Eastern Cooperative Oncology Group (ECOG) Performance status of ≤ 1.
7. Adequate venous access for repeated blood sampling according to the study schedule.
8. Women of child-bearing potential must have a negative serum pregnancy test and agree to remain sexually abstinent, have a partner who is sterile (i.e., vasectomy), or use two medically effective methods of contraception (e.g., oral contraception, barrier methods, spermicide, intrauterine device [IUD]).
9. Able and willing to comply with all study procedures.

Exclusion Criteria:

1. Pregnancy or breastfeeding.
2. History of previous therapeutic HPV vaccination.
3. Prior exposure to an investigational agent or device within 30 days of signing the ICF. Of note, the participant may participate in observational studies.
4. Positive serological test for HIV, Hep B or Hep C or history of HIV infection, Hepatitis B or Hepatitis C (women with cured HCV will be allowed; participant must have had a serologic test performed within 12 months of informed consent).
5. Prior major surgery from which the participant has not yet recovered to baseline.
6. High medical risks because of non-malignant systemic disease or with active uncontrolled infection.
7. Current malignancies at other sites, with the exception of adequately treated basal or squamous cell carcinoma of the skin.
8. Congestive heart failure or prior history of New York Heart Association (NYHA) class III/ IV cardiac disease.
9. Use of topical corticosteroids at or near the intended administration site.
10. Any cardiac pre-excitation syndromes (such as Wolff-Parkinson-White).
11. History of seizures (unless seizure free for 5 years).
12. Tattoos or scars within 2 cm of the intended site of injection or if there is implanted metal within the same limb. Any device implanted in the chest (e.g., cardiac pacemaker or defibrillator) excludes the use of the deltoid muscle on the same side of the body.
13. Active drug or alcohol use or dependence.
14. Imprisonment or compulsory detainment for treatment of either a psychiatric or physical (i.e. infectious disease) illness.
15. History of immunosuppressive or autoimmune disease.
16. Any other illnesses or conditions that in the opinion of the investigator may affect the safety of the participant or limit the evaluation of a participant or any study endpoint.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only female participants with biopsy-proven, Stage IB-IVB inoperable invasive cervical carcinoma associated with HPV-16 and/or HPV-18 were included.
Enrollment: 10 (Actual)
Dates: Start 2014-06-06 (Actual); Primary Completion 2017-09-07 (Actual); Study Completion 2017-09-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Skolnik, MD, Study Director — Inovio Pharmaceuticals
Locations (3):
- United States (3):
  - University of Chicago Medical Center, Chicago, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - Columbia University Medical Center, New York, New York

REFERENCES:
- [Background] Bagarazzi ML, Yan J, Morrow MP, Shen X, Parker RL, Lee JC, Giffear M, Pankhong P, Khan AS, Broderick KE, Knott C, Lin F, Boyer JD, Draghia-Akli R, White CJ, Kim JJ, Weiner DB, Sardesai NY. Immunotherapy against HPV16/18 generates potent TH1 and cytotoxic cellular immune responses. Sci Transl Med. 2012 Oct 10;4(155):155ra138. doi: 10.1126/scitranslmed.3004414. PMID 23052295
- [Background] Diehl MC, Lee JC, Daniels SE, Tebas P, Khan AS, Giffear M, Sardesai NY, Bagarazzi ML. Tolerability of intramuscular and intradermal delivery by CELLECTRA((R)) adaptive constant current electroporation device in healthy volunteers. Hum Vaccin Immunother. 2013 Oct;9(10):2246-52. doi: 10.4161/hv.24702. Epub 2013 Jun 4. PMID 24051434
- See also: Sponsor's Website — http://www.inovio.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Female participants with cervical cancer after chemoradiation for newly diagnosed disease or therapy for recurrent and/or persistent disease were enrolled in 2 study sites between 6th June 2014 to 7th September 2017.
Period: Overall Study
Arm/Group | Cohort I: INO-3112: Curative Intent | Cohort II: INO-3112: Salvage Therapy
Started | 7 | 3
Completed | 6 | 1
Not Completed | 1 | 2
Not completed — Serious Adverse Event | 0 | 1
Not completed — Progression of Disease | 0 | 1
Not completed — Loss of insurance coverage | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort I: INO-3112: Curative Intent | Cohort II: INO-3112: Salvage Therapy | Total
Number analyzed (Participants) | 7 | 3 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.9 (11.63) | 41.7 (14.64) | 46.0 (12.11)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 7 | 3 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 5 | 2 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 5 | 1 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least 1 Treatment Emergent Adverse Event (TEAE)
Description: An adverse event (AE) is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can include any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. A TEAE is any AE either reported for the first time or worsening of a pre-existing event after the first dose of study drug.
Time Frame: Up to 36 weeks
Population: Safety population included all participants who received at least one dose of study treatment plus EP.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort I: INO-3112: Curative Intent | Cohort II: INO-3112: Salvage Therapy
Number analyzed (Participants) | 7 | 3
percentage of participants | 100 [59.0 to 100.0] | 100 [29.2 to 100.0]

2. Primary Outcome: Percentage of Participants With Grade 3 or Higher TEAEs Graded Per Common Terminology Criteria for Adverse Events, Version 4.03 (CTCAE, v 4.03)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can include any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. A TEAE is any AE either reported for the first time or worsening of a pre-existing event after the first dose of study drug. The severity of TEAEs was assessed by the National Cancer Institute's (NCI) Common Terminology Criteria for Adverse Events, version 4.03 (CTCAE,v 4.03). TEAEs were graded on a 5-point scale where 1 = Mild, 2 = Moderate, 3 = Severe, 4 = Potentially life-threatening and 5 = Death.
Time Frame: Up to 36 weeks
Population: Safety population included all participants who received at least one dose of study treatment plus EP.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort I: INO-3112: Curative Intent | Cohort II: INO-3112: Salvage Therapy
Number analyzed (Participants) | 7 | 3
percentage of participants
  Anaemia | 0 [0.0 to 41.0] | 33.3 [0.8 to 90.6]
  Disseminated Intravascular Coagulation | 0 [0.0 to 41.0] | 33.3 [0.8 to 90.6]
  Abdominal Pain | 14.3 [0.4 to 57.9] | 0 [0.0 to 70.8]
  Intestinal Perforation | 0 [0.0 to 41.0] | 33.3 [0.8 to 90.6]
  Pneumonia | 14.3 [0.4 to 57.9] | 0 [0.0 to 70.8]
  Pathological Fracture | 0 [0.0 to 41.0] | 33.3 [0.8 to 90.6]

3. Primary Outcome: Percentage of Participants With Injection Site Reactions
Description: Injection site reactions and administration site pain were evaluated starting 30 minutes following injection/EP. Injection site reactions were assessed in accordance with the 'Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials' (Food and Drug Administration [FDA] Guidance for Industry, September 2007). Local reaction to the injectable product such as pain, tenderness, erythema/redness and induration/swelling were graded on a 4-point scale where: 1 = Mild, 2 = Moderate, 3 = Severe and 4 = Potentially life-threatening.
Time Frame: Up to 36 weeks
Population: Safety population included all participants who received at least one dose of study treatment plus EP.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort I: INO-3112: Curative Intent | Cohort II: INO-3112: Salvage Therapy
Number analyzed (Participants) | 7 | 3
percentage of participants
  Injection Site Bruising | 28.6 [3.7 to 71.0] | 33.3 [0.8 to 90.6]
  Injection Site Discolouration | 0 [0.0 to 41.0] | 33.3 [0.8 to 90.6]
  Injection Site Erythema | 14.3 [0.4 to 57.9] | 0 [0.0 to 70.8]
  Injection Site Haemorrhage | 14.3 [0.4 to 57.9] | 0 [0.0 to 70.8]
  Injection Site Pain | 14.3 [0.4 to 57.9] | 66.7 [9.4 to 99.2]
  Injection Site Swelling | 14.3 [0.4 to 57.9] | 33.3 [0.8 to 90.6]

4. Primary Outcome: Rates of Acute Gastrointestinal, Genitourinary, or Other Chemoradiation Side Effects Above the Expected, Graded Per Acute Radiation Morbidity Scoring Criteria
Time Frame: Up to 36 weeks
Population: The above-mentioned outcome could not be assessed as no data were captured that reflect the expected rates of acute gastrointestinal, genitourinary or other chemoradiation side effects, in order to compare those collected on this study with those from prior studies. While adverse event data related to study therapy were captured, these were not graded per acute radiation morbidity score because of the above-noted limitation. No comparison was thus possible that would reflect rates expected.
Arm/Group | Cohort I: INO-3112: Curative Intent | Cohort II: INO-3112: Salvage Therapy
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Change From Baseline in Hematocrit at the Indicated Time Points
Description: Clinical laboratory parameters (hematology, serum chemistry, and creatine phosphokinase [CPK]) were analyzed using descriptive statistics for actual values and changes from baseline to each study visit.
Time Frame: Baseline and Week 4, 8,12,16,24, 32 and 48
Population: Safety population included all participants who received at least one dose of study treatment plus EP. Number analyzed is the number of participants with data available for analysis at a specified time-point.
Measure: Mean (Standard Deviation); unit: percentage of blood
Arm/Group | Cohort I: INO-3112: Curative Intent | Cohort II: INO-3112: Salvage Therapy
Number analyzed (Participants) | 7 | 3
percentage of blood
  Baseline | 30.87 (3.118) | 35.03 (5.016)
  Change from Baseline at Week 4 | 1.63 (2.553) | -2.10 (2.800)
  Change from Baseline at Week 8: number analyzed (Participants) | 7 | 2
  Change from Baseline at Week 8 | 3.49 (2.805) | -5.90 (6.505)
  Change from Baseline at Week 12: number analyzed (Participants) | 7 | 1
  Change from Baseline at Week 12 | 5.73 (3.722) | 1.60 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  Change from Baseline at Week 16: number analyzed (Participants) | 7 | 1
  Change from Baseline at Week 16 | 5.97 (3.288) | 2.10 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  Change from Baseline at Week 24: number analyzed (Participants) | 1 | 0
  Change from Baseline at Week 24 | 5.10 (NA) — Standard deviation could not be calculated due to insufficient number of participants. |
  Change from Baseline at Week 32: number analyzed (Participants) | 1 | 0
  Change from Baseline at Week 32 | 4.80 (NA) — Standard deviation could not be calculated due to insufficient number of participants. |
  Change from Baseline at Week 48: number analyzed (Participants) | 1 | 0
  Change from Baseline at Week 48 | 4.70 (NA) — Standard deviation could not be calculated due to insufficient number of participants. |

6. Primary Outcome: Change From Baseline in Hemoglobin at the Indicated Time Points
Description: Clinical laboratory parameters (hematology, serum chemistry, creatine phosphokinase [CPK]) were analyzed using descriptive statistics for actual values and changes from baseline to each study visit.
Time Frame: Baseline and Weeks 4, 8,12,16,24, 32 and 48
Population: The safety population included all participants who received at least one dose of study treatment plus EP. Number analyzed is the number of participants with data available for analysis at a specified time-point.
Measure: Mean (Standard Deviation); unit: gram per liter (g/L)
Arm/Group | Cohort I: INO-3112: Curative Intent | Cohort II: INO-3112: Salvage Therapy
Number analyzed (Participants) | 7 | 3
gram per liter (g/L)
  Baseline | 103.29 (10.339) | 112.00 (22.517)
  Change from Baseline at Week 4 | 5.57 (10.048) | -7.00 (9.165)
  Change from Baseline at Week 8: number analyzed (Participants) | 7 | 2
  Change from Baseline at Week 8 | 11.14 (12.402) | -19.00 (24.042)
  Change from Baseline at Week 12: number analyzed (Participants) | 7 | 1
  Change from Baseline at Week 12 | 18.29 (13.889) | 4.00 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  Change from Baseline at Week 16: number analyzed (Participants) | 7 | 1
  Change from Baseline at Week 16 | 20.29 (11.086) | 8.00 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  Change from Baseline at Week 24: number analyzed (Participants) | 1 | 0
  Change from Baseline at Week 24 | 17.00 (NA) — Standard deviation could not be calculated due to insufficient number of participants. |
  Change from Baseline at Week 32: number analyzed (Participants) | 1 | 0
  Change from Baseline at Week 32 | 8.00 (NA) — Standard deviation could not be calculated due to insufficient number of participants. |
  Change from Baseline at Week 48: number analyzed (Participants) | 1 | 0
  Change from Baseline at Week 48 | 7.00 (NA) — Standard deviation could not be calculated due to insufficient number of participants. |

7. Primary Outcome: Change From Baseline in Lymphocytes, Monocytes, Neutrophils and White Blood Cell (WBC) Count at the Indicated Time Points
Description: Clinical laboratory parameters (hematology, serum chemistry, creatine phosphokinase [CPK]) were analyzed using descriptive statistics for actual values and changes from baseline to each study visit. Hematology parameters analyzed for this outcome measure included: white blood cell (WBC) count, count of lymphocytes (L), monocytes (M) and neutrophils (N).
Time Frame: Baseline and Weeks 4, 8,12,16,24, 32 and 48
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: 10^9 cells/liter (10^9/L)
Arm/Group | Cohort I: INO-3112: Curative Intent | Cohort II: INO-3112: Salvage Therapy
Number analyzed (Participants) | 7 | 3
10^9 cells/liter (10^9/L)
  L, Baseline | 0.93 (0.522) | 0.70 (0.400)
  L,Change from Baseline at Week 4 | -0.11 (0.261) | 0.00 (0.200)
  L,Change from Baseline at Week 8: number analyzed (Participants) | 7 | 2
  L,Change from Baseline at Week 8 | -0.04 (0.251) | -0.10 (0.141)
  L, Change from Baseline at Week 12: number analyzed (Participants) | 7 | 1
  L, Change from Baseline at Week 12 | -0.10 (0.283) | -0.20 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  L, Change from Baseline at Week 16: number analyzed (Participants) | 7 | 1
  L, Change from Baseline at Week 16 | 0.01 (0.254) | -0.20 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  L, Change From Baseline at Week 24: number analyzed (Participants) | 1 | 0
  L, Change From Baseline at Week 24 | 0.20 (NA) — Standard deviation could not be calculated due to insufficient number of participants. |
  L, Change from Baseline at Week 32: number analyzed (Participants) | 1 | 0
  L, Change from Baseline at Week 32 | -0.50 (NA) — Standard deviation could not be calculated due to insufficient number of participants. |
  L, Change from Baseline at Week 48: number analyzed (Participants) | 1 | 0
  L, Change from Baseline at Week 48 | -0.40 (NA) — Standard deviation could not be calculated due to insufficient number of participants. |
  M, Baseline | 0.39 (0.121) | 0.30 (0.100)
  M,Change from Baseline at Week 4 | -0.06 (0.172) | 0.07 (0.153)
  M,Change from Baseline at Week 8: number analyzed (Participants) | 7 | 2
  M,Change from Baseline at Week 8 | -0.03 (0.138) | 0.05 (0.212)
  M,Change from Baseline at Week 12: number analyzed (Participants) | 7 | 1
  M,Change from Baseline at Week 12 | -0.03 (0.138) | 0.10 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  M,Change from Baseline at Week 16: number analyzed (Participants) | 7 | 1
  M,Change from Baseline at Week 16 | -0.07 (0.160) | 0.10 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  M,Change from Baseline at Week 24: number analyzed (Participants) | 1 | 0
  M,Change from Baseline at Week 24 | 0.00 (NA) — Standard deviation could not be calculated due to insufficient number of participants. |
  M,Change from Baseline at Week 32: number analyzed (Participants) | 1 | 0
  M,Change from Baseline at Week 32 | -0.40 (NA) — Standard deviation could not be calculated due to insufficient number of participants. |
  M,Change from Baseline at Week 48: number analyzed (Participants) | 1 | 0
  M,Change from Baseline at Week 48 | -0.20 (NA) — Standard deviation could not be calculated due to insufficient number of participants. |
  N, Baseline | 2.60 (2.129) | 4.03 (0.551)
  N,Change from Baseline at Week 4 | 0.43 (0.964) | 0.37 (1.266)
  N,Change from Baseline at Week 8: number analyzed (Participants) | 7 | 2
  N,Change from Baseline at Week 8 | 0.09 (1.188) | 0.85 (0.212)
  N,Change from Baseline at Week 12: number analyzed (Participants) | 7 | 1
  N,Change from Baseline at Week 12 | -0.03 (0.138) | 0.10 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  N,Change from Baseline at Week 16: number analyzed (Participants) | 7 | 1
  N,Change from Baseline at Week 16 | -0.07 (0.160) | 0.10 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  N,Change from Baseline at Week 24: number analyzed (Participants) | 1 | 0
  N,Change from Baseline at Week 24 | 0.00 (NA) — Standard deviation could not be calculated due to insufficient number of participants. |
  N,Change from Baseline at Week 32: number analyzed (Participants) | 1 | 0
  N,Change from Baseline at Week 32 | -0.40 (NA) — Standard deviation could not be calculated due to insufficient number of participants. |
  N,Change from Baseline at Week 48: number analyzed (Participants) | 1 | 0
  N,Change from Baseline at Week 48 | -0.20 (NA) — Standard deviation could not be calculated due to insufficient number of participants. |
  WBC, Baseline | 4.20 (2.239) | 5.30 (0.721)
  WBC, Change from Baseline at Week 4 | 0.33 (0.966) | 0.40 (1.114)
  WBC, Change from Baseline at Week 8: number analyzed (Participants) | 7 | 2
  WBC, Change from Baseline at Week 8 | 0.27 (1.237) | 0.85 (0.212)
  WBC, Change from Baseline at Week 12: number analyzed (Participants) | 7 | 1
  WBC, Change from Baseline at Week 12 | 0.01 (1.771) | 0.40 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  WBC, Change from Baseline at Week 16: number analyzed (Participants) | 7 | 1
  WBC, Change from Baseline at Week 16 | 0.66 (1.279) | 1.40 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  WBC, Change from Baseline at Week 24: number analyzed (Participants) | 1 | 0
  WBC, Change from Baseline at Week 24 | 0.90 (NA) — Standard deviation could not be calculated due to insufficient number of participants. |
  WBC, Change from Baseline at Week 32: number analyzed (Participants) | 1 | 0
  WBC, Change from Baseline at Week 32 | -0.40 (NA) — Standard deviation could not be calculated due to insufficient number of participants. |
  WBC, Change from Baseline at Week 48: number analyzed (Participants) | 1 | 0
  WBC, Change from Baseline at Week 48 | -0.30 (NA) — Standard deviation could not be calculated due to insufficient number of participants. |

8. Primary Outcome: Change From Baseline in Platelet Count at the Indicated Time Points
Description: as for outcome 6
Time Frame: Baseline and Weeks 4,8,12,16,24,32 and 48
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: 10^9 cells/liter (10^9/L)
Arm/Group | Cohort I: INO-3112: Curative Intent | Cohort II: INO-3112: Salvage Therapy
Number analyzed (Participants) | 7 | 3
10^9 cells/liter (10^9/L)
  Platelet Count, Baseline | 259.86 (46.674) | 271.33 (73.704)
  Platelet Count, Change from Baseline at Week 4 | -45.29 (55.479) | 26.00 (48.754)
  Platelet Count, Change from Baseline at Week 8: number analyzed (Participants) | 7 | 2
  Platelet Count, Change from Baseline at Week 8 | -40.57 (39.327) | 93.00 (84.853)
  Platelet Count, Change from Baseline at Week 12: number analyzed (Participants) | 7 | 1
  Platelet Count, Change from Baseline at Week 12 | -41.00 (61.563) | 37.00 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  Platelet Count, Change from Baseline at Week 16: number analyzed (Participants) | 7 | 1
  Platelet Count, Change from Baseline at Week 16 | -32.86 (49.911) | 2.00 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  Platelet Count, Change From Baseline at Week 24: number analyzed (Participants) | 1 | 0
  Platelet Count, Change From Baseline at Week 24 | -17.00 (NA) — Standard deviation could not be calculated due to insufficient number of participants. |
  Platelet Count, Change from Baseline at Week 32: number analyzed (Participants) | 1 | 0
  Platelet Count, Change from Baseline at Week 32 | -68.00 (NA) — Standard deviation could not be calculated due to insufficient number of participants. |
  Platelet Count, Change from Baseline at Week 48: number analyzed (Participants) | 1 | 0
  Platelet Count, Change from Baseline at Week 48 | -73.00 (NA) — Standard deviation could not be calculated due to insufficient number of participants. |

9. Primary Outcome: Change From Baseline in Red Blood Cell (RBC) Count at the Indicated Time Points
Description: as for outcome 6
Time Frame: Baseline and Weeks 4 and 8
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: 10^12 cells/liter
Arm/Group | Cohort I: INO-3112: Curative Intent | Cohort II: INO-3112: Salvage Therapy
Number analyzed (Participants) | 7 | 3
10^12 cells/liter
  RBC Count, Baseline | 3.34 (0.382) | 3.97 (0.586)
  RBC Count, Change from Baseline at Week 4 | 0.07 (0.355) | -0.23 (0.351)
  RBC Count, Change from Baseline at Week 8: number analyzed (Participants) | 7 | 2
  RBC Count, Change from Baseline at Week 8 | 0.23 (0.386) | -0.55 (0.778)

10. Primary Outcome: Change From Baseline in Alkaline Phosphatase, Alanine Aminotransferase, and Aspartate Aminotransferase at the Indicated Time Points
Description: Clinical laboratory parameters (hematology, serum chemistry, creatine phosphokinase [CPK]) were analyzed using descriptive statistics for actual values and changes from baseline to each study visit. Clinical chemistry parameter assessed in this outcome measure included alkaline phosphatase (ALP), alanine amino transferase (ALT) and aspartate amino transferase (AST).
Time Frame: Baseline and Weeks 4,8,12 and 16
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units per liter (U/L)
Arm/Group | Cohort I: INO-3112: Curative Intent | Cohort II: INO-3112: Salvage Therapy
Number analyzed (Participants) | 7 | 3
units per liter (U/L)
  ALP, Baseline | 73.29 (26.606) | 81.33 (10.017)
  ALP, Change from Baseline at Week 4: number analyzed (Participants) | 5 | 3
  ALP, Change from Baseline at Week 4 | 0.20 (13.989) | 14.67 (21.779)
  ALP, Change from Baseline at Week 8: number analyzed (Participants) | 5 | 2
  ALP, Change from Baseline at Week 8 | 3.00 (20.273) | 54.00 (65.054)
  ALP, Change from Baseline at Week 12: number analyzed (Participants) | 5 | 1
  ALP, Change from Baseline at Week 12 | 4.00 (26.448) | 0.00 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  ALP, Change from Baseline at Week 16: number analyzed (Participants) | 5 | 1
  ALP, Change from Baseline at Week 16 | 8.60 (22.233) | 1.00 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  ALT, Baseline | 20.14 (6.793) | 13.00 (9.849)
  ALT, Change from Baseline at Week 4: number analyzed (Participants) | 5 | 3
  ALT, Change from Baseline at Week 4 | 4.60 (13.353) | -3.67 (11.590)
  ALT, Change from Baseline at Week 8: number analyzed (Participants) | 5 | 2
  ALT, Change from Baseline at Week 8 | -5.00 (4.950) | -4.50 (14.849)
  ALT, Change from Baseline at Week 12: number analyzed (Participants) | 5 | 1
  ALT, Change from Baseline at Week 12 | -1.60 (6.229) | -14.00 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  ALT, Change from Baseline at Week 16: number analyzed (Participants) | 5 | 1
  ALT, Change from Baseline at Week 16 | -2.20 (3.768) | -15.00 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  AST, Baseline | 22.71 (6.945) | 17.00 (7.937)
  AST, Change from Baseline at Week 4: number analyzed (Participants) | 5 | 3
  AST, Change from Baseline at Week 4 | 3.20 (8.526) | -5.67 (11.547)
  AST, Change from Baseline at Week 8: number analyzed (Participants) | 5 | 2
  AST, Change from Baseline at Week 8 | -3.80 (6.340) | -5.00 (14.142)
  AST, Change from Baseline at Week 12: number analyzed (Participants) | 5 | 1
  AST, Change from Baseline at Week 12 | 1.20 (13.461) | -15.00 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  AST, Change from Baseline at Week 16: number analyzed (Participants) | 5 | 1
  AST, Change from Baseline at Week 16 | -2.80 (4.658) | -16.00 (NA) — Standard deviation could not be calculated due to insufficient number of participants.

11. Primary Outcome: Change From Baseline in Bicarbonate, Glucose, Blood Urea Nitrogen (BUN), Calcium (Ca), Chloride (Cl), Potassium (K), Magnesium (Mg) and Sodium (Na) at the Indicated Time Points
Description: as for outcome 6
Time Frame: Baseline and Weeks 4,8,12 and 16
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: millimole per liter (mmol/L)
Arm/Group | Cohort I: INO-3112: Curative Intent | Cohort II: INO-3112: Salvage Therapy
Number analyzed (Participants) | 7 | 3
millimole per liter (mmol/L)
  Bicarbonate, Baseline | 25.00 (1.633) | 24.33 (2.082)
  Bicarbonate, Change from Baseline at Week 4: number analyzed (Participants) | 5 | 3
  Bicarbonate, Change from Baseline at Week 4 | 0.00 (1.000) | 3.33 (0.577)
  Bicarbonate, Change from Baseline at Week 8: number analyzed (Participants) | 5 | 2
  Bicarbonate, Change from Baseline at Week 8 | -0.60 (2.074) | 0.00 (2.828)
  Bicarbonate, Change from Baseline at Week 12: number analyzed (Participants) | 5 | 1
  Bicarbonate, Change from Baseline at Week 12 | -1.40 (0.548) | 2.00 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  Bicarbonate, Change from Baseline at Week 16: number analyzed (Participants) | 5 | 1
  Bicarbonate, Change from Baseline at Week 16 | -0.40 (1.140) | 4.00 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  Glucose, Baseline | 6.90 (2.994) | 5.25 (1.042)
  Glucose, Change from Baseline at Week 4: number analyzed (Participants) | 5 | 3
  Glucose, Change from Baseline at Week 4 | -0.60 (0.736) | 1.18 (0.946)
  Glucose, Change from Baseline at Week 8: number analyzed (Participants) | 5 | 2
  Glucose, Change from Baseline at Week 8 | -0.57 (0.839) | 2.69 (2.237)
  Glucose, Change from Baseline at Week 12: number analyzed (Participants) | 5 | 1
  Glucose, Change from Baseline at Week 12 | -0.78 (0.755) | 0.39 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  Glucose, Change from Baseline at Week 16: number analyzed (Participants) | 5 | 1
  Glucose, Change from Baseline at Week 16 | -0.46 (0.308) | -1.44 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  BUN, Baseline | 4.18 (1.897) | 4.17 (1.687)
  BUN, Change from Baseline at Week 4: number analyzed (Participants) | 5 | 3
  BUN, Change from Baseline at Week 4 | 0.86 (1.485) | -1.07 (1.071)
  BUN, Change from Baseline at Week 8: number analyzed (Participants) | 5 | 2
  BUN, Change from Baseline at Week 8 | 0.50 (1.568) | 0.18 (0.757)
  BUN, Change from Baseline at Week 12: number analyzed (Participants) | 5 | 1
  BUN, Change from Baseline at Week 12 | 1.87 (3.085) | -1.79 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  BUN, Change from Baseline at Week 16: number analyzed (Participants) | 5 | 1
  BUN, Change from Baseline at Week 16 | 1.29 (1.686) | -0.71 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  Ca, Baseline | 2.33 (0.089) | 2.37 (0.014)
  Ca, Change from Baseline at Week 4: number analyzed (Participants) | 5 | 3
  Ca, Change from Baseline at Week 4 | 0.05 (0.077) | -0.06 (0.104)
  Ca, Change from Baseline at Week 8: number analyzed (Participants) | 5 | 2
  Ca, Change from Baseline at Week 8 | 0.02 (0.045) | -0.16 (0.088)
  Ca, Change from Baseline at Week 12: number analyzed (Participants) | 5 | 1
  Ca, Change from Baseline at Week 12 | 0.01 (0.086) | -0.08 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  Ca, Change from Baseline at Week 16: number analyzed (Participants) | 5 | 1
  Ca, Change from Baseline at Week 16 | 0.04 (0.121) | -0.15 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  Cl, Baseline | 91.57 (28.757) | 100.00 (3.464)
  Cl, Change from Baseline at Week 4: number analyzed (Participants) | 5 | 3
  Cl, Change from Baseline at Week 4 | 15.40 (34.530) | -1.00 (2.646)
  Cl, Change from Baseline at Week 8: number analyzed (Participants) | 5 | 2
  Cl, Change from Baseline at Week 8 | 14.60 (35.494) | -1.00 (1.414)
  Cl, Change from Baseline at Week 12: number analyzed (Participants) | 5 | 1
  Cl, Change from Baseline at Week 12 | 14.00 (34.785) | 1.00 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  Cl, Change from Baseline at Week 16: number analyzed (Participants) | 5 | 1
  Cl, Change from Baseline at Week 16 | 14.40 (33.923) | 0.00 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  K, Baseline | 4.20 (0.383) | 4.37 (0.252)
  K, Change from Baseline at Week 4: number analyzed (Participants) | 5 | 3
  K, Change from Baseline at Week 4 | -0.16 (0.503) | -0.43 (1.305)
  K, Change from Baseline at Week 8: number analyzed (Participants) | 5 | 2
  K, Change from Baseline at Week 8 | -0.06 (0.391) | -0.65 (1.061)
  K, Change from Baseline at Week 12: number analyzed (Participants) | 5 | 1
  K, Change from Baseline at Week 12 | -0.02 (0.466) | -0.70 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  K, Change from Baseline at Week 16: number analyzed (Participants) | 5 | 1
  K, Change from Baseline at Week 16 | -0.14 (0.365) | -1.00 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  Mg, Baseline: number analyzed (Participants) | 1 | 0
  Mg, Baseline | 0.41 (NA) — Standard deviation could not be calculated due to insufficient number of participants. |
  Na, Baseline | 141.29 (3.147) | 138.67 (1.528)
  Na, Change from Baseline at Week 4: number analyzed (Participants) | 5 | 3
  Na, Change from Baseline at Week 4 | 0.00 (2.915) | 1.67 (4.726)
  Na, Change from Baseline at Week 8: number analyzed (Participants) | 5 | 2
  Na, Change from Baseline at Week 8 | -0.20 (1.924) | -0.50 (3.536)
  Na, Change from Baseline at Week 12: number analyzed (Participants) | 5 | 1
  Na, Change from Baseline at Week 12 | -1.20 (2.280) | 4.00 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  Na, Change from Baseline at Week 16: number analyzed (Participants) | 5 | 1
  Na, Change from Baseline at Week 16 | -0.60 (1.517) | 3.00 (NA) — Standard deviation could not be calculated due to insufficient number of participants.

12. Primary Outcome: Change From Baseline in Albumin and Total Protein at the Indicated Time Points
Description: as for outcome 6
Time Frame: Baseline and Weeks 4,8,12 and 16
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: grams per liter (g/L)
Arm/Group | Cohort I: INO-3112: Curative Intent | Cohort II: INO-3112: Salvage Therapy
Number analyzed (Participants) | 7 | 3
grams per liter (g/L)
  Albumin, Baseline | 42.00 (2.000) | 40.33 (3.215)
  Albumin, Change from Baseline at Week 4: number analyzed (Participants) | 5 | 3
  Albumin, Change from Baseline at Week 4 | -1.00 (1.000) | -1.00 (1.000)
  Albumin, Change from Baseline at Week 8: number analyzed (Participants) | 5 | 2
  Albumin, Change from Baseline at Week 8 | 0.80 (1.304) | -2.50 (3.536)
  Albumin, Change from Baseline at Week 12: number analyzed (Participants) | 5 | 1
  Albumin, Change from Baseline at Week 12 | 0.60 (2.191) | -2.00 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  Albumin, Change from Baseline at Week 16: number analyzed (Participants) | 5 | 1
  Albumin, Change from Baseline at Week 16 | 1.00 (1.871) | -1.00 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  Total protein, Baseline | 68.86 (4.488) | 73.67 (3.215)
  Total protein, Change from Baseline at Week 4: number analyzed (Participants) | 5 | 3
  Total protein, Change from Baseline at Week 4 | 1.20 (2.168) | -2.67 (3.215)
  Total protein, Change from Baseline at Week 8: number analyzed (Participants) | 5 | 2
  Total protein, Change from Baseline at Week 8 | 2.80 (4.087) | -5.50 (3.536)
  Total protein, Change from Baseline at Week 12: number analyzed (Participants) | 5 | 1
  Total protein, Change from Baseline at Week 12 | 2.20 (5.805) | -2.00 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  Total protein, Change from Baseline at Week 16: number analyzed (Participants) | 5 | 1
  Total protein, Change from Baseline at Week 16 | 3.20 (5.357) | -2.00 (NA) — Standard deviation could not be calculated due to insufficient number of participants.

13. Primary Outcome: Change From Baseline in Creatine Phosphokinase (CPK) at the Indicated Time Points
Description: as for outcome 6
Time Frame: Baseline and Week 16
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units per liter (U/L)
Arm/Group | Cohort I: INO-3112: Curative Intent | Cohort II: INO-3112: Salvage Therapy
Number analyzed (Participants) | 7 | 3
units per liter (U/L)
  CPK, Baseline | 46.9 (9.30) | 42.7 (15.50)
  CPK, Change from Baseline at Week 16: number analyzed (Participants) | 5 | 1
  CPK, Change from Baseline at Week 16 | 18.8 (15.80) | 30.0 (NA) — Standard deviation could not be calculated due to insufficient number of participants.

14. Primary Outcome: Change From Baseline in Creatinine and Total Bilirubin at the Indicated Time Points
Description: as for outcome 6
Time Frame: Baseline and Weeks 4, 8,12 and 16
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: micromoles per liter (umol/L)
Arm/Group | Cohort I: INO-3112: Curative Intent | Cohort II: INO-3112: Salvage Therapy
Number analyzed (Participants) | 7 | 3
micromoles per liter (umol/L)
  Creatinine, Baseline | 66.93 (16.817) | 70.72 (8.840)
  Creatinine, Change from Baseline at Week 4: number analyzed (Participants) | 5 | 3
  Creatinine, Change from Baseline at Week 4 | 5.83 (7.543) | 2.95 (5.104)
  Creatinine, Change from Baseline at Week 8: number analyzed (Participants) | 5 | 2
  Creatinine, Change from Baseline at Week 8 | -1.59 (7.193) | 8.84 (12.502)
  Creatinine, Change from Baseline at Week 12: number analyzed (Participants) | 5 | 1
  Creatinine, Change from Baseline at Week 12 | 6.01 (8.442) | -17.68 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  Creatinine, Change from Baseline at Week 16: number analyzed (Participants) | 5 | 1
  Creatinine, Change from Baseline at Week 16 | 3.36 (8.015) | -8.84 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  Total Bilirubin, Baseline | 7.82 (4.922) | 6.84 (4.524)
  Total Bilirubin, Change from Baseline at Week 4: number analyzed (Participants) | 5 | 3
  Total Bilirubin, Change from Baseline at Week 4 | -1.71 (4.837) | -1.71 (2.962)
  Total Bilirubin, Change from Baseline at Week 8: number analyzed (Participants) | 5 | 2
  Total Bilirubin, Change from Baseline at Week 8 | -1.37 (4.083) | -1.71 (4.837)
  Total Bilirubin, Change from Baseline at Week 12: number analyzed (Participants) | 5 | 1
  Total Bilirubin, Change from Baseline at Week 12 | -1.03 (5.353) | 0.00 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  Total Bilirubin, Change from Baseline at Week 16: number analyzed (Participants) | 5 | 1
  Total Bilirubin, Change from Baseline at Week 16 | -0.00 (6.283) | 0.00 (NA) — Standard deviation could not be calculated due to insufficient number of participants.

15. Secondary Outcome: Change From Baseline in the Combined HPV-16 and HPV-18 E6 and E7 Antigen Specific Spot-Forming Units Per Million Peripheral Blood Mononuclear Cell (SFU/10^6 PBMC)
Description: Whole blood and serum samples to be tested for antibodies to the human papillomavirus (HPV) E6 and E7 proteins and/or T-lymphocytes producing interferon-gamma (IFN-γ) elicited by INO-3112 were assessed by enzyme-linked immunosorbent spot-forming assay (ELISpot).
Time Frame: Baseline and Weeks 2, 4, 6, 8, 10,12,14,16, 24, 32, 36, 40 and 48
Population: Modified intention-to-treat (mITT) population included all participants receiving at least one study treatment plus EP as assigned. Number analyzed is the number of participants with data available for analysis at a specified time-point.
Measure: Mean (Standard Deviation); unit: SFU/10^6 PBMC
Arm/Group | Cohort I: INO-3112: Curative Intent | Cohort II: INO-3112: Salvage Therapy
Number analyzed (Participants) | 7 | 3
SFU/10^6 PBMC
  Baseline: number analyzed (Participants) | 3 | 3
  Baseline | 8.6 (6.03) | 6.7 (2.89)
  Increase from Baseline at Week 2: number analyzed (Participants) | 0 | 2
  Increase from Baseline at Week 2 |  | 1.7 (2.35)
  Increase from Baseline at Week 4: number analyzed (Participants) | 3 | 2
  Increase from Baseline at Week 4 | 26.4 (29.84) | 2.5 (3.54)
  Increase from Baseline at Week 6: number analyzed (Participants) | 1 | 2
  Increase from Baseline at Week 6 | 20.0 (NA) — Standard deviation could not be calculated due to insufficient number of participants. | 24.2 (12.96)
  Increase from Baseline at Week 8: number analyzed (Participants) | 2 | 2
  Increase from Baseline at Week 8 | 68.3 (49.50) | 0.0 (0.0)
  Increase from Baseline at Week 10: number analyzed (Participants) | 2 | 0
  Increase from Baseline at Week 10 | 50.0 (21.21) |
  Increase from Baseline at Week 12: number analyzed (Participants) | 3 | 1
  Increase from Baseline at Week 12 | 353.3 (472.30) | 6.7 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  Increase from Baseline at Week 14: number analyzed (Participants) | 2 | 0
  Increase from Baseline at Week 14 | 27.5 (8.24) |
  Increase from Baseline at Week 16: number analyzed (Participants) | 3 | 1
  Increase from Baseline at Week 16 | 310.3 (460.00) | 53.3 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  Increase from Baseline at Week 24: number analyzed (Participants) | 3 | 0
  Increase from Baseline at Week 24 | 244.2 (324.77) |
  Increase from Baseline at Week 32: number analyzed (Participants) | 3 | 1
  Increase from Baseline at Week 32 | 121.9 (133.43) | 10.0 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  Increase from Baseline at Week 36: number analyzed (Participants) | 1 | 0
  Increase from Baseline at Week 36 | 6.7 (NA) — Standard deviation could not be calculated due to insufficient number of participants. |
  Increase from Baseline at Week 40: number analyzed (Participants) | 2 | 0
  Increase from Baseline at Week 40 | 246.3 (341.18) |
  Increase from Baseline at Week 48: number analyzed (Participants) | 2 | 0
  Increase from Baseline at Week 48 | 248.8 (351.79) |

16. Secondary Outcome: E6 Antigen Specific Anti-HPV-16/18 Antibody Titers Assessed by Enzyme-linked Immunosorbent Assay (ELISA)
Description: Antigen-specific humoral responses against HPV E6 and E7 antigens induced by INO-3112 were measured using ELISA. Commercially available recombinant human HPV-16 and HPV-18 proteins were used to assess the induction of binding antibodies to each of the antigen components.
Time Frame: Baseline and Weeks 2, 4, 6, 8, 10,12,14,16, 24, 32, 36, 40 and 48
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: log titer
Arm/Group | Cohort I: INO-3112: Curative Intent | Cohort II: INO-3112: Salvage Therapy
Number analyzed (Participants) | 7 | 3
log titer
  HPV-16 ,Baseline | 0.0 (0.00) | 0.0 (0.00)
  HPV-16, Week 2: number analyzed (Participants) | 2 | 2
  HPV-16, Week 2 | 2.5 (3.54) | 0.0 (0.00)
  HPV-16, Week 4: number analyzed (Participants) | 6 | 3
  HPV-16, Week 4 | 0.7 (1.60) | 0.0 (0.00)
  HPV-16, Week 6: number analyzed (Participants) | 2 | 2
  HPV-16, Week 6 | 2.5 (3.54) | 0.0 (0.00)
  HPV-16, Week 8: number analyzed (Participants) | 7 | 2
  HPV-16, Week 8 | 0.6 (1.48) | 0.0 (0.00)
  HPV-16, Week 10: number analyzed (Participants) | 3 | 1
  HPV-16, Week 10 | 0.0 (0.00) | 0.00 (NA) — Standard deviation could not be calculated due to an insufficient number of participants.
  HPV-16, Week 12: number analyzed (Participants) | 5 | 1
  HPV-16, Week 12 | 0.8 (1.75) | 0.0 (NA) — Standard deviation could not be calculated due to an insufficient number of participants.
  HPV-16, Week 14: number analyzed (Participants) | 2 | 0
  HPV-16, Week 14 | 2.0 (2.77) |
  HPV-16, Week 16: number analyzed (Participants) | 7 | 1
  HPV-16, Week 16 | 1.4 (2.44) | 0.0 (NA) — Standard deviation could not be calculated due to an insufficient number of participants.
  HPV-16, Week 24: number analyzed (Participants) | 6 | 1
  HPV-16, Week 24 | 3.0 (2.36) | 0.0 (NA) — Standard deviation could not be calculated due to an insufficient number of participants.
  HPV-16, Week 32: number analyzed (Participants) | 6 | 1
  HPV-16, Week 32 | 1.7 (2.59) | 0.0 (NA) — Standard deviation could not be calculated due to an insufficient number of participants.
  HPV-16, Week 36: number analyzed (Participants) | 4 | 1
  HPV-16, Week 36 | 0.0 (0.00) | 0.0 (NA) — Standard deviation could not be calculated due to an insufficient number of participants.
  HPV-16, Week 40: number analyzed (Participants) | 3 | 0
  HPV-16, Week 40 | 3.3 (2.89) |
  HPV-16, Week 48: number analyzed (Participants) | 3 | 0
  HPV-16, Week 48 | 3.7 (3.26) |
  HPV-18, Baseline | 0.0 (0.00) | 0.0 (0.00)
  HPV-18, Week 2: number analyzed (Participants) | 2 | 2
  HPV-18, Week 2 | 3.1 (4.32) | 0.0 (0.00)
  HPV-18, Week 4: number analyzed (Participants) | 6 | 3
  HPV-18, Week 4 | 0.7 (1.60) | 0.0 (0.00)
  HPV-18, Week 6: number analyzed (Participants) | 2 | 2
  HPV-18, Week 6 | 0.0 (0.00) | 0.0 (0.00)
  HPV-18, Week 8: number analyzed (Participants) | 7 | 2
  HPV-18, Week 8 | 0.6 (1.48) | 0.0 (0.00)
  HPV-18, Week 10: number analyzed (Participants) | 3 | 1
  HPV-18, Week 10 | 1.3 (2.26) | 0.0 (NA) — Standard deviation could not be calculated due to an insufficient number of participants
  HPV-18, Week 12: number analyzed (Participants) | 5 | 1
  HPV-18, Week 12 | 0.8 (1.75) | 6.1 (NA) — Standard deviation could not be calculated due to an insufficient number of participants.
  HPV-18, Week 14: number analyzed (Participants) | 2 | 0
  HPV-18, Week 14 | 0.0 (0.00) |
  HPV-18, Week 16: number analyzed (Participants) | 7 | 1
  HPV-18, Week 16 | 1.4 (2.53) | 6.1 (NA) — Standard deviation could not be calculated due to an insufficient number of participants.
  HPV-18, Week 24: number analyzed (Participants) | 6 | 1
  HPV-18, Week 24 | 0.7 (1.60) | 0.0 (NA) — Standard deviation could not be calculated due to an insufficient number of participants.
  HPV-18, Week 32: number analyzed (Participants) | 6 | 1
  HPV-18, Week 32 | 1.3 (2.02) | 0.0 (NA) — Standard deviation could not be calculated due to an insufficient number of participants.
  HPV-18, Week 36: number analyzed (Participants) | 4 | 1
  HPV-18, Week 36 | 1.5 (3.05) | 0.0 (NA) — Standard deviation could not be calculated due to an insufficient number of participants.
  HPV-18, Week 40: number analyzed (Participants) | 3 | 0
  HPV-18, Week 40 | 1.3 (2.26) |
  HPV-18, Week 48: number analyzed (Participants) | 3 | 0
  HPV-18, Week 48 | 0.0 (0.00) |

17. Secondary Outcome: E7 Antigen Specific Anti-HPV-16/18 Antibody Titers Assessed by ELISA
Description: as for outcome 16
Time Frame: Baseline and Weeks 2, 4, 6, 8, 10, 12, 14, 16, 24, 32, 36, 40 and 48
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: log titer
Arm/Group | Cohort I: INO-3112: Curative Intent | Cohort II: INO-3112: Salvage Therapy
Number analyzed (Participants) | 7 | 3
log titer
  HPV-16, Baseline | 0.0 (0.00) | 0.0 (0.00)
  HPV-16, Week 2: number analyzed (Participants) | 3 | 2
  HPV-16, Week 2 | 0.0 (0.00) | 2.0 (2.77)
  HPV-16, Week 4: number analyzed (Participants) | 6 | 3
  HPV-16, Week 4 | 0.7 (1.60) | 0.0 (0.00)
  HPV-16, Week 6: number analyzed (Participants) | 2 | 2
  HPV-16, Week 6 | 0.0 (0.00) | 0.0 (0.00)
  HPV-16, Week 8: number analyzed (Participants) | 6 | 2
  HPV-16, Week 8 | 0.8 (2.05) | 3.6 (5.10)
  HPV-16, Week 10: number analyzed (Participants) | 3 | 1
  HPV-16, Week 10 | 3.3 (3.09) | 7.2 (NA) — Standard deviation could not be calculated due to an insufficient number of participants.
  HPV-16, Week 12: number analyzed (Participants) | 5 | 1
  HPV-16, Week 12 | 2.0 (2.85) | 7.2 (NA) — Standard deviation could not be calculated due to an insufficient number of participants.
  HPV-16, Week 14: number analyzed (Participants) | 2 | 0
  HPV-16, Week 14 | 3.1 (4.32) |
  HPV-16, Week 16: number analyzed (Participants) | 7 | 1
  HPV-16, Week 16 | 2.1 (2.75) | 7.2 (NA) — Standard deviation could not be calculated due to an insufficient number of participants.
  HPV-16, Week 24: number analyzed (Participants) | 6 | 1
  HPV-16, Week 24 | 2.7 (3.13) | 7.2 (NA) — Standard deviation could not be calculated due to an insufficient number of participants.
  HPV-16, Week 32: number analyzed (Participants) | 6 | 1
  HPV-16, Week 32 | 2.1 (2.38) | 7.2 (NA) — Standard deviation could not be calculated due to an insufficient number of participants.
  HPV-16, Week 36: number analyzed (Participants) | 5 | 1
  HPV-16, Week 36 | 1.6 (2.14) | 0.0 (NA) — Standard deviation could not be calculated due to an insufficient number of participants.
  HPV-16, Week 40: number analyzed (Participants) | 3 | 0
  HPV-16, Week 40 | 0.0 (0.00) |
  HPV-16, Week 48: number analyzed (Participants) | 2 | 0
  HPV-16, Week 48 | 0.0 (0.00) |
  HPV-18, Baseline | 0.0 (0.00) | 0.0 (0.00)
  HPV-18, Week 2: number analyzed (Participants) | 3 | 2
  HPV-18, Week 2 | 1.7 (2.89) | 0.0 (0.00)
  HPV-18, Week 4: number analyzed (Participants) | 6 | 3
  HPV-18, Week 4 | 0.8 (2.05) | 0.0 (0.00)
  HPV-18, Week 6: number analyzed (Participants) | 2 | 2
  HPV-18, Week 6 | 5.0 (1.55) | 0.0 (0.00)
  HPV-18, Week 8: number analyzed (Participants) | 6 | 2
  HPV-18, Week 8 | 2.4 (3.72) | 0.0 (0.00)
  HPV-18, Week 10: number analyzed (Participants) | 3 | 1
  HPV-18, Week 10 | 1.3 (2.26) | 0.0 (NA) — Standard deviation could not be calculated due to an insufficient number of participants.
  HPV-18, Week 12: number analyzed (Participants) | 5 | 1
  HPV-18, Week 12 | 2.2 (3.26) | 7.2 (NA) — Standard deviation could not be calculated due to an insufficient number of participants.
  HPV-18, Week 14: number analyzed (Participants) | 2 | 0
  HPV-18, Week 14 | 2.0 (2.77) |
  HPV-18, Week 16: number analyzed (Participants) | 7 | 1
  HPV-18, Week 16 | 3.5 (3.56) | 7.2 (NA) — Standard deviation could not be calculated due to an insufficient number of participants.
  HPV-18, Week 24: number analyzed (Participants) | 6 | 1
  HPV-18, Week 24 | 1.2 (2.94) | 8.3 (NA) — Standard deviation could not be calculated due to an insufficient number of participants.
  HPV-18, Week 32: number analyzed (Participants) | 6 | 1
  HPV-18, Week 32 | 1.9 (3.05) | 8.3 (NA) — Standard deviation could not be calculated due to an insufficient number of participants.
  HPV-18, Week 36: number analyzed (Participants) | 5 | 1
  HPV-18, Week 36 | 0.0 (0.00) | 8.3 (NA) — Standard deviation could not be calculated due to an insufficient number of participants.
  HPV-18, Week 40: number analyzed (Participants) | 3 | 0
  HPV-18, Week 40 | 5.2 (4.51) |
  HPV-18, Week 48: number analyzed (Participants) | 2 | 0
  HPV-18, Week 48 | 3.6 (5.10) |

ADVERSE EVENTS:
Time Frame: Up to 36 weeks
Arm/Group | Cohort I: INO-3112: Curative Intent | Cohort II: INO-3112: Salvage Therapy
All-Cause Mortality (participants affected / at risk) | 0/7 | 1/3
Serious Adverse Events (participants affected / at risk) | 3/7 | 2/3
Other Adverse Events (participants affected / at risk) | 7/7 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort I: INO-3112: Curative Intent (N=7) | Cohort II: INO-3112: Salvage Therapy (N=3)
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Intestinal Perforation (Gastrointestinal disorders) | 0 | 1
Endometritis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort I: INO-3112: Curative Intent (N=7) | Cohort II: INO-3112: Salvage Therapy (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Tachycardia (Cardiac disorders) | 2 | 1
Ear Pain (Ear and labyrinth disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Abdominal Pain Lower (Gastrointestinal disorders) | 1 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Defaecation Urgency (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 0
Dry Mouth (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Motility Disorder (Gastrointestinal disorders) | 1 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 2 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Hiatus Hernia (Gastrointestinal disorders) | 1 | 0
Large Intestine Polyp (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 3 | 1
Rectal Ulcer (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2
Chest Pain (General disorders) | 1 | 0
Fatigue (General disorders) | 2 | 0
Injection Site Bruising (General disorders) | 2 | 1
Injection Site Discolouration (General disorders) | 0 | 1
Injection Site Erythema (General disorders) | 1 | 0
Injection Site Haemorrhage (General disorders) | 1 | 0
Injection Site Pain (General disorders) | 1 | 2
Injection Site Swelling (General disorders) | 1 | 1
Malaise (General disorders) | 1 | 0
Peripheral Swelling (General disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Hepatic Steatosis (Hepatobiliary disorders) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Pyometra (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 1
Ligament Sprain (Injury, poisoning and procedural complications) | 1 | 0
Radiation Proctopathy (Injury, poisoning and procedural complications) | 0 | 1
Weight Decreased (Investigations) | 2 | 0
White Blood Cell Count Decreased (Investigations) | 1 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 2 | 1
Pain In Jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1
Dysgeusia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 0
Neuropathy Peripheral (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Parosmia (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 1
Insomnia (Psychiatric disorders) | 2 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Nocturia (Renal and urinary disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
Urge Incontinence (Renal and urinary disorders) | 1 | 0
Urinary Incontinence (Renal and urinary disorders) | 2 | 0
Coital Bleeding (Reproductive system and breast disorders) | 1 | 0
Dyspareunia (Reproductive system and breast disorders) | 1 | 0
Uterine Pain (Reproductive system and breast disorders) | 1 | 0
Uterine Prolapse (Reproductive system and breast disorders) | 1 | 0
Vaginal Haemorrhage (Reproductive system and breast disorders) | 2 | 0
Vaginal Stricture (Reproductive system and breast disorders) | 0 | 1
Vulvovaginal Pain (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Excessive Granulation Tissue (Skin and subcutaneous tissue disorders) | 1 | 0
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 1
Hot Flush (Vascular disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-27): https://cdn.clinicaltrials.gov/large-docs/11/NCT02172911/Prot_SAP_000.pdf